CLINICAL TRIAL: NCT05000437
Title: The Effectiveness and Safety of High Intensity Interval Training Based on Oxidative Stress and Inflammatory Markers in the Management of Overweight Male Subjects
Brief Title: The Effectiveness and Safety of HIIT in Overweight Male Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Indonesia University (Other)
Responsible Party: Principal Investigator, Nani Cahyani Sudarsono, Head of Sports Medicine Study Program, Indonesia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 20-09-1081
Record Dates: First submitted 2021-05-29; First posted 2021-08-11 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Overweight; Overweight or Obesity
Keywords: high intensity interval training; overweight; young male
MeSH Terms: conditions — Overweight; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- High Intensity Interval Training (Experimental): single arm intervention, with high intensity interval training
  Interventions: Other: HIIT

INTERVENTIONS:
Other: HIIT — 3x/week high intensity interval training for 12 weeks

SUMMARY:
Increased prevalence of overweight and obesity is one of the main health problems recently. Energy balance from nutrition intake and energy expenditure through physical activity, especially structured physical activity, is needed to prevent overweight individuals become obese individuals. This research objective is to explore the effectiveness and safety of structured high intensity interval training in male young adults subjects with overweight based on change of body composition, oxidative stress and inflammatory markers. This research used experimental model to test structured high intensity interval training program with pre-post test in single group. Comprehensive analysis of training effect in this research consists of measurement of several parameters, such as body composition, inflammatory markers, and oxidative stress markers as the benchmark of training safety. Browning white adipose tissue and cognitive function are complement parameters to the assessment of training effectiveness. Daily food record and physical activity for 3 x 24 hours will be carried out periodically to control confounding factors.

DETAILED DESCRIPTION:
* Subjects are recruited via e-flyer distributed online across university departments. Individual who is interested in study participation fills out screening form. Research assistants screen subjects eligibility. Subjects are coded based on the order of screening form fulfillment.
* Research assistants are using the standard operational procedures for each assessments. Training for the research assistants precedes the data collection to ensure the similarity of understanding and skills during measurements. One research assistant responsible for scheduling the assessments and training sessions. Continuous evaluation are planned weekly to provide room for improvements in the process of data collection.
* Sample size assessment is measured from 5 primary output by a research assistants using sample size calculation website for single intervention clinical trial.
* Investigator use paper based data collection for each assessment and during training sessions. Subject are encouraged to report any symptoms and signs during intervention period in each meeting with the research assistants or via online messaging. Any reports will be documented in separated form. One research assistant makes sure the data fields are completed in each measurements and during training sessions. The assistant also check the similarity of the data entered in the master table.
* Data analysis will be lead by one research assistant using newest version of SPSS software. The analysis will be started after the baseline measurement is completed although the data collection is not finished. All numeric data will be presented as mean and standard deviations if normally distributed or median and minimum maximum range if not normally distributed. Paired t-test will be used to identify the difference before and after the intervention if the data are normally distributed. If the data are not normally distributed, Wilcoxon test will be used to identify the difference before and after the intervention.

To ensure that there is no missing data, the research assistant who responsible for data completeness will perform daily checking. Any missing data will be stated and immediately completed. Research assistants will provide close supervision for each subject to ensure the delivery of all necessary reports.

ELIGIBILITY:
Inclusion Criteria:

* overweight (BMI 25 - 29,9)
* live in Jakarta and greater area
* willing to participate

Exclusion Criteria:

* smoking
* any medical health problems (epilepsy, cardiovascular disease, kidney and liver problems, history of fractures, tendon and ligament injuries)

Ages: 18 Years to 30 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2020-11-01 (Actual); Primary Completion 2021-10-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
cardiorespiratory fitness | 12 weeks
  VO2Max in ml/kg/minute
body mass index | week 4
  weight and height combined as BMI in kg/m2
body mass index | week 8
  weight and height combined as BMI in kg/m2
body mass index | week 12
  weight and height combined as BMI in kg/m2
body fat mass | week 4
  total fat mass in the body as percentage
body fat mass | week 8
  total fat mass in the body as percentage
body fat mass | week 12
  total fat mass in the body as percentage
visceral fat | week 4
  body fat stored within abdominal cavity as ratings
visceral fat | week 8
  body fat stored within abdominal cavity as ratings
visceral fat | week 12
  body fat stored within abdominal cavity as ratings
waist circumference | week 4
  circumference measured in the horizontal plane midway between the lowest ribs and the iliac crest as cm
waist circumference | week 8
  circumference measured in the horizontal plane midway between the lowest ribs and the iliac crest as cm
waist circumference | week 12
  circumference measured in the horizontal plane midway between the lowest ribs and the iliac crest as cm
lipid profile | 12 weeks
  total cholesterol, HDL cholesterol, LDL cholesterol, triglyceride
antioxidant level | 12 weeks
  SOD in U/mg
free radicals level | 12 weeks
  MDA in nmol/mg
inflammation | 12 weeks
  TNF-alpha in microgram/ml
interleukin level | 12 weeks
  IL-6 nanogram/ml

SECONDARY OUTCOMES:
Fat Burning Effect | week 1, 6, 12
  FGF21
Myokin | week 1, 6, 12
  Irisin
Cognitive Function Screening | week 1 and 12
  Montreal Cognitive Assessment as score
Working memory Capacity | week 1 and 12
  N-Back test as percentage of correct answers
Executive Function | week 1 and 12
  Trail Making Test A and B as seconds

CONTACTS AND LOCATIONS:
Overall Officials: Nani Sudarsono, Principal Investigator — Fakultas Kedokteran Universitas Indonesia
Locations (2):
- Indonesia (2):
  - Fakultas Kedokteran Universitas Indonesia, Jakarta Pusat, DKI Jakarta
  - Universitas Indonesia, Jakarta Pusat, DKI Jakarta

DOCUMENTS (1):
  • Study Protocol, Statistical Analysis Plan, and Informed Consent Form (2021-10-08): https://cdn.clinicaltrials.gov/large-docs/37/NCT05000437/Prot_SAP_ICF_001.pdf